CLINICAL TRIAL: NCT03165071
Title: A Single-center, Open Label, Single-dose Study to Investigate the Effect of Severe Renal Impairment on the Pharmacokinetics of ACT-132577
Brief Title: A Study to Evaluate ACT-132577 in Healthy Subjects and in People With Severe Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AC-080-105; 2016-005077-12 (EudraCT Number)
Record Dates: First submitted 2017-05-23; First posted 2017-05-24 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Severe Renal Impairment; Healthy Subjects
MeSH Terms: conditions — Renal Insufficiency | interventions — aprocitentan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ACT-132577 (50 mg) (Experimental): 8 healthy subjects and 8 subjects with severe renal function impairment will receive a single oral dose of 50 mg ACT-132577 administered as capsule following an overnight fast
  Interventions: Drug: ACT-132577

INTERVENTIONS:
Drug: ACT-132577 — Capsule
  Other Names: Aprocitentan

SUMMARY:
The primary purpose of this study is to investigate the fate of ACT-132577 in healthy subjects and in people with severe kidney disease

ELIGIBILITY:
Inclusion Criteria:

ALL SUBJECTS:

* Signed informed consent in the local language prior to any study-mandated procedure;
* Male/female aged 18 to 65 years (inclusive) at screening;
* Body mass index of 18.0 to 32.0 kg/m2 (inclusive) at screening. Body weight at least 50 kg;
* Women of childbearing potential must have a negative serum pregnancy test and use reliable birth controls up to 30 days after the end of study treatment.

HEALTHY SUBJECTS:

* Normal renal function confirmed by the estimated glomerular filtration rate (eGFR) determined at screening;
* Healthy on the basis of physical examination, cardiovascular assessments and laboratory tests.

SEVERE RENAL FUNCTION IMPAIRMENT SUBJECTS:

- Severe renal function impairment is defined by eGFR estimated at screening between 15 mL/min/1.73 m2 and 29 mL/min/1.73 m2 (inclusive).

Exclusion Criteria:

ALL SUBJECTS:

* Pregnant or lactating women;
* Known hypersensitivity to ACT-132577 or drugs of the same class, or any of their excipients;
* Known hypersensitivity or allergy to natural rubber latex;
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

SEVERE RENAL FUNCTION IMPAIRMENT SUBJECTS:

* End-stage renal disease that requires dialysis;
* Hemoglobin concentration < 9 g/dL;
* History of severe renal stenosis;
* Serum potassium concentration > 5.5 mmol/L;
* Presence of severe cardiac disease;
* History of clinically relevant bleeding disorder;
* Presence of any organ disorder, with the exception of renal function impairment, or use of any medication which might interfere with the pharmacokinetics of ACT-132577;
* Known life-threatening disease with a life expectancy of less than 1 year;
* Presence of unstable diabetes mellitus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-06-03 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of ACT-132577 | From baseline to up to 16 days
  Cmax of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profiles
Area under the plasma concentration-time curves during a dosing interval [AUC(0-t)] of ACT-132577 | From baseline to up to 16 days
  AUC(0-T) of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profiles
Area under the plasma concentration-time curves from time 0 to inf [AUC(0-inf)] | From baseline to up to 16 days
  AUC(0-inf) of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profiles

SECONDARY OUTCOMES:
Time to reach Cmax (tmax) of ACT-132577 | From baseline to up to 16 days
  tmax of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profiles
Terminal half-life [t(1/2)] | From baseline to up to 16 days
  t1/2 of ACT-132577 will be derived by non-compartmental analysis of the plasma concentration-time profiles
Incidence of treatment-emergent adverse events | From baseline to up to 16 days
  The percentage of subjects with treatment-emergent adverse events will be reported
Incidence of adverse events leading to premature discontinuation of study treatment | From baseline to up to 16 days
  The number of subjects who prematurely discontinued the study treatment due to an adverse event will be reported
Incidence of any clinical relevant findings in ECG variables | From baseline to up to 16 days
  The number of subjects with any treatment-emergent electrocardiogram (ECG) abnormalities will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA, Pilsen, Czechia

REFERENCES:
- [Background] Sidharta PN, Ulc I, Dingemanse J. Single-Dose Pharmacokinetics and Tolerability of Aprocitentan, a Dual Endothelin Receptor Antagonist, in Subjects with Severe Renal Function Impairment. Clin Drug Investig. 2019 Nov;39(11):1117-1123. doi: 10.1007/s40261-019-00837-x. PMID 31435905